CLINICAL TRIAL: NCT05704036
Title: Estrogen Supplementation and Bone Health in Women With CF (STURDY)
Brief Title: Estrogen Supplementation and Bone Health in Women With CF
Acronym: STURDY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00307525
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis; Hypoestrogenism
Keywords: Bone Mineral Density; Osteoporosis; Young Adult; Adolescent; Premenopause; Estradiol; Bone Disease; Bone Diseases, Metabolic; Hormones; Quality of Life
MeSH Terms: conditions — Cystic Fibrosis; Osteoporosis; Bone Diseases; Bone Diseases, Metabolic | interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Observational Study (No Intervention): Participants will complete three study visits (baseline, 6 months, and 12 months) involving DXAs (bone density assessment), x-rays, blood draws, and questionnaires.
- Transdermal Estradiol/Cyclic Progesterone (Experimental): Participants will apply transdermal estradiol patches (0.1 mg/day) weekly for 12 months following baseline study visits. Participants not already using a progesterone-containing contraceptive will also take progesterone (200 mg) for 10 days per month.
  Interventions: Drug: Transdermal estrogen; Drug: Progesterone

INTERVENTIONS:
Drug: Transdermal estrogen — Transdermal estradiol 0.1 mg/day, applied once weekly
  Other Names: Transdermal estradiol; Climara
  Arms: Transdermal Estradiol/Cyclic Progesterone
Drug: Progesterone — Progesterone 200 mg daily for 10 days/month, if participant is not on progesterone-containing contraceptive
  Other Names: Prometrium
  Arms: Transdermal Estradiol/Cyclic Progesterone

SUMMARY:
The goal of this study is to learn about the role of estrogen and other hormones in bone development in adolescent and young adult women with cystic fibrosis (CF). The study has two main components, an observational study and a feasibility sub-study. The main questions it aims to answer are:

* How do different forms of hormonal contraception (e.g. birth control pill or other progesterone only methods) impact bone health?
* Is a study of transdermal estradiol (estrogen skin patches) feasible in this group?
* How does transdermal estradiol impact bone health and quality of life?

Participants in the observational study will have three study visits (baseline, 6 months, and 12 months). At all visits, participants will have blood drawn and will complete questionnaires. At the baseline and 12 month visits, participants will additionally have x-rays and DXAs (bone density assessment). Between visits, participants will complete brief questionnaires. Researchers will compare various measurements over time to assess the impact of different forms of hormonal contraception.

Participants in the feasibility sub-study will apply transdermal estradiol patches once weekly for 12 months, fill out brief quality-of-life surveys in between study visits, and complete blood draws and questionnaires at four study visits (baseline, 3 months, 6 months, and 12 months). The participants will also have x-rays and DXAs performed at the baseline and 12 month visits. Researchers will examine changes in various measurements to determine the impact of transdermal estradiol.

ELIGIBILITY:
Observational Study:

Inclusion Criteria:

* CF Diagnosis
* Females who have had at least 1 menstrual cycle
* Planning to use same formulation of estrogen supplementation (or none) for duration of study

Exclusion Criteria:

* Use of anti-osteoporosis therapy including anti-resorptives such as bisphosphonates or anabolic agents such as teriparatide or denosumab
* Conditions in which bone loss is known to be present or expected to occur, such as lactation
* Pregnant or planning to become pregnant
* In the opinion of the CF care team or study investigators participant should not participate in the study
* Inability to provide informed consent/assent

Feasibility Sub-Study:

Inclusion Criteria:

* All of above and
* <35 years old
* At least 2 years after first menstrual cycle
* Symptoms of low estrogen and/or low serum estradiol levels (< 50 pg/mL)

Exclusion Criteria:

* All of above and
* Contraindications to transdermal estradiol
* Current use of systemic estrogen (such as estrogen-containing oral contraceptive pill)
* Previous lung or liver transplant
* Use of chronic systemic glucocorticoids
* Severe vitamin D deficiency (serum 25(OH)D < 6 ng/mL)
* Conditions increasing risk of clot: history of previous deep vein thrombus or pulmonary embolism, current immobility, current peripherally inserted central catheter or mediport, known hypercoagulable condition
* Baseline study visit falls between 1 and 8 weeks after initiation of CF transmembrane receptor (CFTR) modulator
* Currently in pulmonary exacerbation
* Recent antibiotic use within the past 4 weeks for an acute pulmonary exacerbation
* Unwilling or unable to use a non-estrogen containing method of contraception such as barrier, abstinence, or progesterone-only method

Ages: 0 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in lumbar spine bone mineral density assessed by dual-energy x-ray absorptiometry (DXA) | Baseline and 12 months

SECONDARY OUTCOMES:
Change in serum procollagen type I intact N-terminal propeptide (P1NP) levels (mcg/L) | Baseline and 12 months
  P1NP is a marker of bone turnover.
Change in serum C-terminal telopeptide of type I collagen (CTX-1) levels (pg/mL) | Baseline and 12 months
  CTX-1 is a marker of bone turnover.
Change in quality of life as assessed by Cystic Fibrosis Respiratory Symptom Diary - Chronic Respiratory Infection Symptom Score (CFRSD-CRISS) questionnaire | Baseline and 12 months
  CFRSD-CRISS is a brief survey to assess quality of life of people with cystic fibrosis that will be taken by participants twice per month. The questionnaire is scored from 0-100 with higher scores indicating increased symptom severity.

OTHER OUTCOMES:
Study procedure completion rate | Evaluated at completion of study, approximately two years
  Percentage of participants enrolled in study who complete all study procedures.
Acceptability as determined by participant report | Across 12 months of study participation per participant
  Acceptability during study participation by 5 point Likert scale, with a score or 3 or greater considered acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Malinda Wu, MD, MSc, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No